CLINICAL TRIAL: NCT04577261
Title: A Prospective Study To Evaluate The FEMORAL NECK SYSTEM (FNS) In The Treatment Of INTRA-CAPSULAR FEMORAL Neck Fractures
Brief Title: FNS (FEMORAL NECK SYSTEM) Study
Acronym: FNS
Status: Active, not recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00066583
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Femoral Neck Fractures
Keywords: neck fractures; implant failure; osteotomy
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Femoral Neck System (FNS) Participants: Participants who will undergo surgery to treat a fractured femoral neck using the FNS (Femoral Neck System)

SUMMARY:
A post-market, prospective study to evaluate the reoperation rate of displaced and nondisplaced femoral neck fractures treated with the Femoral Neck System (FNS)™

DETAILED DESCRIPTION:
To evaluate the re-operation rate for any reason of displaced and non-displaced femoral neck fractures treated with the Femoral Neck System (FNS)™ at one year post-operation. The Femoral Neck System (FNS)™ represents a new generation of implants designed to improve outcomes in the treatment of femoral neck fractures. These implants offer a fixed angle construct and all of its mechanical advantages with regards to neutralizing shear and providing stability while not exerting a rotational malreduction force on the fracture. The FNS system has been shown to compare favorably to traditional fixed angle constructs in a cadaveric model

ELIGIBILITY:
Inclusion Criteria:

* The subject must provide written informed consent
* The subject must be eighteen (18) years of age or older.
* The subject must be willing and able to make all required study visits including one (1) year post-operative follow-up.
* The subject must be able to follow instructions.
* Subject has experienced displaced or non-displaced intracapsular femoral neck fracture

Exclusion Criteria:

* Subject with fracture occurring more than 7 days prior to the date of surgery
* Subject has more than one fracture on target extremity.
* Subject is obese as defined by a Body Mass Index (BMI) > 45 at the time of surgery.
* Subject, in the opinion of the Investigator, has an emotional or neurological condition that preludes cooperation and compliance with the rehabilitation regimen.
* Therapy with another investigational agent within thirty (30) days of Screening or planned therapy with another investigational agent during the course of the study.
* Subject has a physical condition that, in the opinion of the Investigator, would preclude adequate implant support or impede healing (e.g. blood supply impairment insufficient bone quality or quantity, or an active, local or systemic infection). If this is identified at the time of surgery, the subject will be screen failed.
* Subject has undergone previous surgery on the target hip.
* Current systemic therapy with cytotoxic drugs.
* Subjects with a history of poor compliance with medical treatment.
* Subjects with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject has experienced displaced or non-displaced intracapsular femoral neck fracture
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Re-operation rate | Year 1 post-operation
  Re-operation rate for any reason of displaced and non-displaced femoral neck fractures treated with the Femoral Neck System (FNS)™

SECONDARY OUTCOMES:
Timed Up and Go (TUG) time | Week 6, Months 3, 6, and 12
  The Timed Up and Go Test assesses mobility, balance, walking ability, and fall risk in adults by measuring time, in seconds, that it takes the individual to stand from a chair, walk a distance of 10 feet, walk back to the chair, and sit down. The subject will perform the test in their everyday footwear with their walking aid (cane, walker), if applicable. Normal healthy elderly usually complete the task in ten seconds or less. Very frail or weak elderly with poor mobility may take 2 minutes or more. 8
European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) Score | Baseline, Week 6, Months 3, 6, and 12
  The EuroQol EQ-5D-5L is a standardized instrument for use as a measurement of health outcome. It consists of a descriptive system with 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), which are each assigned five levels (no problems, slight problems, moderate problems, severe problems and extreme problems) The first part (descriptive system with 5 dimensions) is scored using the Health state index scores. Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility.
European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) - VAS (Visual Analogue Scale) Score | Baseline, Week 6, Months 3, 6, and 12
  The EuroQol EQ-5D-5L is a standardized instrument for use as a measurement of health outcome. It consists of a descriptive system with 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), which are each assigned five levels (no problems, slight problems, moderate problems, severe problems and extreme problems), as well as, a Visual Analogue Scale where subjects indicate a numerical value from 0-100 where 0 is the worst imaginable health state and 100 is the best imaginable health state.
Visual Analogue Scale (VAS) for Pain Score | Baseline, Week 6, Months 3, 6, and 12
  The Visual Analogue Scale is simply a line of fixed length, on which the subject marks their experience of pain with a single stroke of a pen - The subject will record their level of pain on a 100 mm visual analog scale - the scale will be marked 'no pain' on the left side of the scale and 'severe pain' at the right end of the scale - It is generally accepted that a pain VAS score of 30, 70, and 100 indicates the upper boundaries of mild, moderate, and severe pain intensity
Number of Participants with Quality of Fracture Reduction | Baseline, Week 6, Months 3, 6, and 12
  Appropriate reduction will be defined as the principal compressive trabeculae measuring >160° in the AP view and <5° of posterior angulation in the lateral view. If reduction is acceptable in both views, it will be classified as grade I. Grade II will be indicative of one plane of malreduction, and grade III will be indicative of malreduction in both radiographic views.
  Pre-operative radiographs will be reviewed and classified as displaced (e.g. Garden III & IV) or non-displaced (e.g. Garden I & II) femoral neck fractures by the Investigator at each site Pauwel Classification (Type I - 30 degrees, Type II - 50 degrees, Type III - 70 degrees)
Active Straight Leg Raise (ASLR) Assessment Score | Baseline, Week 6, Months 3, 6, and 12
  The ALSR assessment provides information about the ability of load transfer and motor control strategies in the lumbo/pelvic/hip complex. ASLR will be performed with the subject in a relaxed supine position with legs straight and feet apart. Subjects will be instructed to raise their operated leg 20cm above the examination table without bending the knee and without pelvic movement relative to the trunk. A score will be provided by the subject for the operated limb on a six-point Likert scale (0 = not difficult at all, 1 = minimally difficult; 2 = somewhat able to do, 3 = fairly difficult, 4 = very difficult, 5 = unable to do) -Lower score denotes better outcome
Number of Participants with Intraoperative complications | Baseline, Week 6, Months 3, 6, and 12
  Number of Participants with Intraoperative complications
Radiographic outcomes including quality of fracture reduction | Baseline, Week 6, Months 3, 6, and 12
  Perform radiology imaging collecting both anteroposterior (AP) and lateral images of the target hip to ensure the FNS is properly implanted - (healed, non-union, aligned, mal-union, osteonecrosis of femoral head, no osteonecrosis of femoral head, none)
Number of Construct failure past 6 months | Months 6 and 12
  Construct failure past typical femoral neck fracture healing period (past 6 months)
Time to return to full weight-bearing | Week 6, Months 3, 6, and 12
  Time to return to full weight-bearing
Ambulatory status from pre-injury to study completion | Baseline, Week 6, Months 3, 6, and 12
  Subjects will be assessed as "Unaided", "Using a cane", "Using a walker" or "Bed to Chair"
Length of hospital stay | Week 6, Months 3, 6, and 12
  Length of hospital stay
Number of Hospital readmission for any reason | Week 6, Months 3, 6, and 12
  Number of Hospital readmission for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Eben A Carroll, MD, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kenan S, Gold A, Salai M, Steinberg E, Ankory R, Chechik O. Long-Term Outcomes Following Reduction and Fixation of Displaced Subcapital Hip Fractures in the Young Elderly. Isr Med Assoc J. 2015 Jun;17(6):341-5. PMID 26233991
- [Background] Han S, Oh M, Yoon S, Kim J, Kim JW, Chang JS, Ryu JS. Risk Stratification for Avascular Necrosis of the Femoral Head After Internal Fixation of Femoral Neck Fractures by Post-Operative Bone SPECT/CT. Nucl Med Mol Imaging. 2017 Mar;51(1):49-57. doi: 10.1007/s13139-016-0443-8. Epub 2016 Aug 11. PMID 28250858
- [Background] Farooq MA, Orkazai SH, Okusanya O, Devitt AT. Intracapsular fractures of the femoral neck in younger patients. Ir J Med Sci. 2005 Oct-Dec;174(4):42-5. doi: 10.1007/BF03168981. PMID 16445160
- [Background] Campenfeldt P, Hedstrom M, Ekstrom W, Al-Ani AN. Good functional outcome but not regained health related quality of life in the majority of 20-69 years old patients with femoral neck fracture treated with internal fixation: A prospective 2-year follow-up study of 182 patients. Injury. 2017 Dec;48(12):2744-2753. doi: 10.1016/j.injury.2017.10.028. Epub 2017 Oct 18. PMID 29106948